CLINICAL TRIAL: NCT04153838
Title: Estimating Premorbid Intellectual Functioning in the Paediatric Population and Developing a Reliable Means for Quantifying Abnormal Change in Cognitive Functions as Children Develop
Brief Title: Estimating Premorbid Intellectual Functioning in Children and Measuring Change in Cognitive Functioning as Children Develop
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-064-19
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Cognitive Impairment
Keywords: Neuropsychology
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children: A group of 'typically' developing children (aged between 6 years and 16 years 11 months) from the general paediatric population will be recruited; with the sample distributed evenly across 6 age bands (i.e. ages 6-7 years, 8-9 years, 10-11 years, 12-13 years, 14-15 years, and 16 years+).
  Interventions: Other: Cognitive test administration

INTERVENTIONS:
Other: Cognitive test administration — Specifically chosen cognitive tests will be administered to all participants twice; with an approximate 12 month gap between initial testing and follow-up testing.

SUMMARY:
Diagnosing and documenting the presence of abnormal change in cognitive functions (such as reasoning abilities) in children over time is of upmost importance when it comes to evaluating the impact of neurological injury, disease, and interventions designed to help improve wellbeing. Unfortunately however, current methods for detecting cognitive impairment and monitoring for abnormal cognitive change in children over time are seriously flawed. By assessing typically developing children's cognitive functioning at two different time points, this study intends to generate new normative data that will significantly improve measurement accuracy when it comes to evaluating the impact of neurological injury and disease on a child's cognitive abilities.

DETAILED DESCRIPTION:
Neurological injury and disease can substantially affect how children's brains work. This can severely impair cognitive abilities and general development. On a day-to-day level, completing everyday tasks, socialising successfully with peers, and getting on with school work can become much more difficult than it was before.

Helpfully, supports and treatments are available that can reduce the negative effects of neurological impairment on a child's cognitive functioning in order to maximise developmental outcomes. However, to deliver appropriate interventions, we must correctly estimate the impact of injury or illness on cognitive abilities and accurately measure how successful treatments are at improving outcomes. Unfortunately, reliable ways of doing this simply do not exist at this time. Consequently, accurate disease (effects) monitoring is seriously undermined; potentially compromising a child's medical management and, thereby, future developmental outcomes.

This study intends to addresses this grave shortcoming by developing reliable ways of measuring the cognitive effects of neurological disease or injury at diagnosis and beyond. Of note, by providing a mechanism to better inform clinical/medical management decisions, completion of this study will help contribute to health and social care aims of enabling children to realise their developmental potential.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be aged between 6 years 0 months and 16 years 11 months 364 days
* Participants must be enrolled into a local mainstream school and have English as their first language
* Participants must not have sustained a previous brain-injury and not suffer from any other neurological illness (please see exclusion criteria below)

Exclusion Criteria:

* Individuals born significantly premature, that have a diagnosis of learning disability, a known neurological illness, or who have had a previous head-injury that required hospitalisation will be excluded from taking part in the study
* Individuals with a current mental health problem for which they are receiving treatment or those with substance misuse problems will also be excluded
* Participants unable to give informed consent will likewise be excluded

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A group of schoolchildren (aged between 6 years and 16 years 11 months) from the general paediatric population will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Obtained intelligence quotient (IQ) score | Baseline
  A child's obtained Full Scale IQ score from a standardised assessment of intelligence constitutes the main outcome variable for this study
Change in obtained intelligence quotient (IQ) score (at 12 month follow-up) | 12 months
  A child's obtained Full Scale IQ score at 12 months follow-up also constitutes a main outcome variable for this study

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Downey, Principal Investigator — NHS Grampian
Locations (1):
- Royal Aberdeen Children's Hospital, Aberdeen, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No